CLINICAL TRIAL: NCT03024554
Title: Evaluation of Safety and Efficacy of the Bifurcated Multilayer Flow Modulator (BMFM®).
Acronym: STREAMLINER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiatis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-2013
Record Dates: First submitted 2017-01-05; First posted 2017-01-19 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2019-07

CONDITIONS: Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal
Keywords: aortic aneurysm involving iliac arteries; abdominal aortic aneurysm; MFM; Multilayer Flow Modulator; Multilayer Stent
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): aortic aneurysm involving iliac arteries treatment with the Bifurcated Multilayer Flow Modulator (BMFM)
  Interventions: Device: Implantation of the Bifurcated Multilayer Flow Modulator

INTERVENTIONS:
Device: Implantation of the Bifurcated Multilayer Flow Modulator
  Other Names: BMFM; BMFM kit

SUMMARY:
To determine the safety and efficacy of the BMFM® kit in the use for the endovascular treatment of aortic aneurysms involving iliac arteries. The BMFM® kit is an adaptation of the aortic MFM® to the aortoiliac bifurcation morphology. It should be noted that the aortic MFM® has CE mark approval for the aortic aneurysm treatment.

DETAILED DESCRIPTION:
Endovascular approaches to TAAAs have evolved during the past decade. The initial experiences with fenestrated and branched endografts have shown that total endovascular repair is effective and may reduce morbidity rates in patients with arch, thoracoabdominal and pararenal aneurysms.

The Cleveland Clinic group has recently reported on their updated clinical experience with the first 633 patients treated by fenestrated and branched endografts. Operative mortality was 1.8% for pararenal, 5.2% for types I to III, and 2.3% for type IV TAAAs .

However, 30-40% of TAAA patients remain unsuitable for EVAR due to unfavorable proximal neck anatomy. There is also an increased incidence of type I proximal endoleak when established f-EVAR guidelines are disregarded, often leading to endovascular re-intervention or surgical conversion.

Currently, the use of the bifurcated stent-graft for the infrarenal aneurysm involving iliac arteries treatment has received wide distribution. The application of endovascular technology to treat infrarenal aneurysm is now commonplace because the implantation of an infrarenal endoprosthesis is a relatively simple procedure requiring adequately long proximal seal zone, diameter measurements and accurate longitudinal device placement. However, designing and implanting a device, which will accommodate the visceral branches, is more complex.

The infrarenal with unfavorable or insufficient proximal neck as well as juxtarenal aneurysms, which involve iliac arteries, could be treated by combination of the Fenestrated Stent Graft with the Bifurcated Stent Graft.

The principal limitation of this technology is the customized nature of fenestrated stent-graft design. From planning to delivery, the process may take in excess of 6 weeks, which restricts the application of f-EVAR to stable elective patients. This procedure is complex, costly and the implantation time is quite long. It must be conducted in expert centers with sophisticated infrastructure (hybrid room). Preservation of visceral aortic branches requires precise graft construction and deployment.

There are reports in the literature of emergent f-EVAR, but the success of these procedures relies on on-site modification of commercially available endografts.

Until an "off-the-shelf'' device is designed to be compatible with the majority of patients, ''off-label'' surgeon-modified devices remain the only option in emergencies when open repair is prohibited. The "off-the-shelf" devices are likely to allow treatment of more than 60% to 80% of patients with complex aneurysms but these standardized designs have not yet been tested clinically in large number of patients with long follow-up In the absence of widely available endografts designs, a number of centers have reported creative techniques to incorporate the visceral arteries, such as "chimney", "sandwich" , "octopus" , "periscope" and physician-modified endografts. However, these approaches are limited by off-label indications, lack of quality control, violation of basic engineering concepts and questionable durability.

One of the drawbacks linked to the use of parallel endografts (mainly for the "chimney technique") remains the imperfect seal inherent to this technique. This side by side configuration leads to gutter along the parallel endografts, which can result in type I endoleaks between the main body of the graft and branched grafts; "Gutter endoleaks" continuously pressurize the aneurysm. The gutters between the main aortic graft, the chimney graft (GC), and the aortic wall should be as narrow as possible to avoid endoleaks, which can be harmful and -almost always- require re-intervention.

Thoraco Abdominal Aneurysms involving iliac arteries remain a challenge for EVAR. Dilatation of the common iliac artery (CIA) often leaves no distal landing zone for commercially available stent grafts, which have a maximum diameter of 28 mm. Furthermore, aneurysms extended to the internal iliac artery (IIA) make endovascular repair even more difficult.

A common method allowing endovascular treatment of these aneurysms is occlusion of the IIA, thereby creating a distal landing zone in the external iliac artery (EIA). However, sacrificing the pelvic blood flow while occluding the internal iliac artery often results in buttock claudication and impotence, as well as other complications such as colonic infarction, gut or spinal cord ischemia. The frequency of these complications varies between 13% and 55% and they can impair quality of life substantially.

Successful treatment of aortoiliac aneurysms involves branch vessel preservation and long-term protection from rupture. While EVAR has totally eclipsed open surgery because of its lower mortality and morbidities, the durability of EVAR can be questioned because of the need for re-intervention and incidence of late aneurysm-related complications . Notably, long-term failure can arise because of the loss of proper seal at the proximal or distal landing zone of the stent-graft (type I endoleaks). Importantly, common iliac diameter can be considered as a predictor of late sac enlargement, as well as implantation outside Manufacturer's Instructions For Use (IFU). Furthermore, Benharash et al. managed to demonstrate that iliac fixation is of high importance for the prevention of device migration, regardless of proximal attachment type.

Iliac artery involvement incidence in abdominal aortic aneurysms (AAAs) is estimated at 20 to 30 %. Hence, nearly a third of all patients presenting with AAAs for repair might not fit within the IFU for standard EVAR device based on iliac diameters. A common approach to ensure appropriate landing zone for iliac components of endografts involves extension into the external iliac artery, with or without concomitant hypogastric artery embolization and coverage. While unilateral coiling has been demonstrated to have relatively low rates of complication, occlusion of the hypogastric artery due to stent graft placement can lead to major complications, as mentioned above. Given the significant morbidity associated with these complications, industry has developed branch technology for hypogastric preservation.

The Multilayer Flow Modulator (MFM®) provides a less complex interventional approach for aortic aneurysm treatment. This device is an uncovered, self-expanding wire mesh with high radial force and flexibility. It is designed to modulate blood-flow dynamics by relieving local peak wall shear stress (PWSS), achieving stabilization of aneurysm-sac or false lumen pressure and preserving side-branch patency.

The clinical benefits of this technology have been assessed and shown in case reports and clinical studies of thoracoabdominal aneurysm, type B dissection, pararenal aortic aneurysm and peripheral artery aneurysm (celiac, hepatic, renal, iliac, subclavian) (48-79). Also the prospective multicenter registry of peripheral and visceral aneurysms (69) and the prospective multicenter STRATO Trial of TAAA (78), show good results at 12-month follow-up.

The MFM® eliminates flow vortex pressure and laminates the outside the device along the aneurysm wall in the same direction of the blood stream. Laminated flow possess unique and protective effects on endothelial cells as well as the ability to promote thrombus progressive formation within the aneurysmal sac. The MFM® addresses not only those issues in a very unique fashion, providing a uniform interface between the artery wall and the blood flow, but its favorable compliance means the device will not be subjected to the same drag forces a conventional stent graft will undergo..

Laminating the blood flow within the aneurysm, promoting thrombus formation within the aneurysmal sac and re-establishing a favorable biochemical and biomechanical balance of endothelial homeostasis, the MFM® addresses aneurysm related issues and outcomes in a novel manner. With aneurysmal stabilization and thrombosis, the MFM® excludes the aneurysm from the circulation rather physically and physiologically than mechanically, as other conventional grafts do. Thanks to the intrinsic porosity of the device, branches are kept patent and well perfused, thus abolishing the risk for collaterals occlusion and consequent ischemia.

STREAMLINER study is an international, multicentre, prospective, non-randomized study. It is designed to evaluate the safety and efficacy of BMFM® kit use. Approximately 40 patients, from up to 12 centres in Europe, Israel, Morocco, Bahrain and Turkey, will be enrolled and screened per the protocol-required inclusion, exclusion criteria, in order to obtain 30 completed patients. The results will be compared with published results for other treatment modalities in the literature. Patients will be included only after obtaining fully informed consent, after conducting all pre-operative examinations required, with respect for all inclusion and exclusion criteria. For early demonstration of efficacy and safety an interim analysis will be performed after the 10 first enrolled patients will complete their 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

* Age over 18
* Life expectancy > 12 months
* Aortic aneurysms involving iliac arteries
* Healthy proximal and distal landing zone
* Adequate arterial access
* Healthy branches and collaterals (no stenosis or previously treated by angioplasty)
* Informed consent understood, signed and patient agrees to all follow-up visits

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

* Aneurysm rupture, impending or contained rupture
* Aortic dissection
* Aortic root aneurysm
* Pleural effusion
* Prior all surgical procedure within 30 days unless procedure is in preparation for device implantation or planned within 30 days post stent deployment
* Myocardial infarction or cerebral vascular accident within 6 weeks of treatment
* Presence/suspicion of connective tissue disorders, for example, Marfan or Ehlers-Danlos etc.
* Contraindications to the anticoagulant or/ and antiplatelet medications
* Allergic reaction to a contrast agent
* Patient with undergoing or planned chemotherapy
* History of bleeding disorder (coagulopathy) or thrombophilia
* Shaggy aorta
* Takayasu's arteritis
* Presence/suspicion of infection (for example: mycotic aorta)
* The use of the MFM® with stent-grafts or previously implanted stent-grafts
* Pregnant or breastfeeding woman
* Patients included in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with unruptured aneurysm | 12 months
  the prevention of aortic aneurysm rupture by the BMFM, in stabilizing it, will be evaluated with the number of patient presenting with unruptured aneurysm at the specified timepoint.
Mortality 30 days, 6 months and 1 year aneurysm-related | 30 days, 6 months and 12 months

SECONDARY OUTCOMES:
Number of branches and collaterals patent | 12 months
  The patency of branches will be evaluated as follows: the number of branches patent will be evaluated on the total number of branches covered by the device (baseline data)
Mortality 30 days, 6 months and 1 year not aneurysm-related | 30 days, 6 months and 12 months
Number of Major Adverse Events | 12 months
  Number of patients with Major Adverse Evens
Technical success | The technical success is evaluated/recorded post-procedure and presented in the 12 months report.
  successful delivery and deployment of the BMFM® kit
Procedural/in-hospital evaluations (Anesthesia time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  descriptive statistics on Anesthesia time (min)
Procedural/in-hospital evaluations (Fluoroscopy time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on fluoroscopy time (min)procedure time; time to hospital discharge
Procedural/in-hospital evaluations (Constrast Volume) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on contrast product volume (ml)
Procedural/in-hospital evaluations (Estimated Blood loss) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on contrast Estimated Blood loss (ml)
Procedural/in-hospital evaluations (procedure time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on procedure time (min); time to hospital discharge
Procedural/in-hospital evaluations (time to hospital discharge) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on time to hospital discharge (days).

CONTACTS AND LOCATIONS:
Locations (7):
- Hôpitaux IRIS Sud Molière Longchamps, Brussels, Uccle, Belgium
- City Hospital Clinic, Sofia, Bulgaria
- CMC Coeur et Vaisseaux, Salé, Morocco
- Romania (2):
  - ELYTIS Hospital: Spital Multidisciplinar şi Policlinică, Iași
  - European Hospital Polisano, Sibiu
- Slovenia (2):
  - University Medical Centre Ljubljana, Ljubljana
  - Maribor University Medical Centre, Maribor

IPD SHARING:
Plan to Share IPD: No